CLINICAL TRIAL: NCT05102383
Title: Evaluation of Wear Experience With a Water Surface Daily Disposable Contact Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Jennifer Fogt, Associate Professor of Clinical Optometry, Ohio State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2021H0305
Record Dates: First submitted 2021-10-15; First posted 2021-11-01 (Actual); Results first posted 2023-12-06 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Contact Lens

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- All participants (Experimental): All participants have habitual Comfilcon A Toric lenses optimized for wear over 2 weeks. Then all participants are fit with the Verofilcon A study daily disposable lenses with water surface treatment for astigmatism.
  Interventions: Device: Comfilcon A Toric contact lenses; Device: Verofilcon A for Astigmatism Daily Disposable contact lenses

INTERVENTIONS:
Device: Comfilcon A Toric contact lenses — Monthly replacement contact lenses
Device: Verofilcon A for Astigmatism Daily Disposable contact lenses — Daily disposable contact lenses

SUMMARY:
The purpose of this study is to assess the wear experience of existing wearers of a monthly replacement contact lens after they have been fit with a daily disposable contact lens that has water surface treatment.

ELIGIBILITY:
Inclusion Criteria:

* Must be a current wearer of Comfilcon A contact lenses
* Distance visual acuity of 20/25 or better with current contact lenses
* Good general health (defined by medication use that has not changed within the last month and the absence of medical conditions or treatments that are deemed confounding to the data as determined by the PI)
* Ability to give informed consent
* Willing to spend time for the study, which includes attending three study visits and be willing to wear contact lenses on days between study visits.
* Either gender.
* Any racial or ethnic origin.

Exclusion Criteria:

* No current ocular inflammation or infection.
* Not currently pregnant or lactating

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2022-04-19 (Actual); Study Completion 2022-04-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Fogt, OD MS, Principal Investigator — The Ohio State University College of Optometry
Locations (1):
- The Ohio State University College of Optometry, Columbus, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Habitual Lens Optimization Followed by Refitting With Study Lenses: All participants are re-fit with habitual Biofinity Toric lenses to optimize vision. Lenses were worn for 2 weeks before returning to be refit with daily disposable lenses with water surface treatment.
Period: Overall Study
Arm/Group | Habitual Lens Optimization Followed by Refitting With Study Lenses
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Habitual Lens Optimization Followed by Refitting With Study Lenses
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.2 (4.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 7
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 19
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Subjective Assessment of Overall Comfort With Verofilcon A Daily Disposable Lenses for Astigmatism
Description: Participants will complete a Visual Analog Scale survey of overall comfort (0-100 Scale with 0 anchored with "Poor Comfort" and 100 anchored as "Excellent Comfort")
Time Frame: 3 weeks
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Habitual Lens Optimization Followed by Refitting With Study Lenses
Number analyzed (Participants) | 30
units on a scale | 91 [80 to 100]

ADVERSE EVENTS:
Time Frame: 1 month
Groups:
- All Participants: All participants are re-fit to optimize fit and vision with their habitual Comfilcon A lenses before being fit with the study lenses. These optimized lenses were worn for 2 weeks before returning to be refit with the study daily disposable lenses.
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 1/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=30)
Hordeolum/Stye (Eye disorders) | 1 (30) — A hordeolum (eyelid bump) occurred during the course of the study while wearing the study lens, used warm compresses to treat, then resumed study lens wear and completed the study. Participant reported historical hordeola before participation also.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2021-07-08): https://cdn.clinicaltrials.gov/large-docs/83/NCT05102383/Prot_002.pdf